CLINICAL TRIAL: NCT07237880
Title: Use of Papaverine to Shorten the Second Stage/Duration of Labor in Pregnant Women After Cervical Ripening by Double-balloon Catheter
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0100-24-HYMC
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Labor, Induced
MeSH Terms: interventions — Papaverine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm Name: Papaverine (Experimental): "Participants receive 80 mg intravenous papaverine immediately after removal of the double-balloon catheter, together with initiation of oxytocin augmentation."
  Interventions: Drug: Papaverine 80 mg IV
- Arm Type: Placebo Comparator (Placebo Comparator): "Participants receive intravenous normal saline immediately after removal of the double-balloon catheter, together with initiation of oxytocin augmentation."
  Interventions: Drug: Placebo (Normal Saline)

INTERVENTIONS:
Drug: Papaverine 80 mg IV — Single intravenous dose of 80 mg papaverine administered immediately after removal of the double-balloon cervical ripening catheter. The medication is given by the midwife as part of the randomized, double-blind protocol, followed by initiation of oxytocin augmentation according to standard labor management.
  Arms: Arm Name: Papaverine
Drug: Placebo (Normal Saline) — Single intravenous dose of normal saline administered immediately after removal of the double-balloon cervical ripening catheter. The placebo is administered in an identical manner to the papaverine intervention as part of the randomized, double-blind protocol, followed by initiation of oxytocin augmentation.
  Arms: Arm Type: Placebo Comparator

SUMMARY:
This prospective, randomized, double-blind controlled trial aims to evaluate whether intravenous papaverine, administered immediately after the removal of a double-balloon catheter used for cervical ripening, can shorten the duration of labor in term pregnant women undergoing induction of labor. Papaverine is an antispasmodic medication that relaxes smooth muscle and is commonly used in obstetrics, although its effect on labor progression following mechanical cervical ripening has not been fully studied.

Eligible participants include nulliparous and multiparous women with a singleton pregnancy at 37-42 weeks, admitted for induction of labor with a double-balloon catheter. After catheter removal, participants will be randomized in a 1:1 ratio to receive either 80 mg intravenous papaverine or placebo (normal saline), administered by the midwife who is not involved in clinical decision-making. Clinical staff and participants will remain blinded to group allocation.

The primary outcomes are the time from drug administration to complete cervical dilation and the duration of the second stage of labor. Secondary outcomes include mode of delivery, maternal complications (such as perineal tears and postpartum hemorrhage), oxytocin augmentation duration and maximum dose, and neonatal outcomes.

This study seeks to determine whether papaverine can safely and effectively reduce labor duration following mechanical cervical ripening.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant individuals aged 18-50 years
* Singleton pregnancy
* Gestational age 37-42 weeks
* Admission for induction of labor with a double-balloon catheter
* Planned vaginal delivery
* Ability to provide informed consent

Exclusion Criteria:

* Previous cesarean delivery
* Multiple gestation
* Contraindication to vaginal delivery
* Known hypersensitivity to papaverine
* Known major fetal anomaly
* Any condition requiring immediate delivery or precluding safe participation (as determined by the treating physician)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — "Only pregnant individuals who identify as female are eligible to participate. The study population consists exclusively of pregnant women admitted for induction of labor at term."
Enrollment: 184 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2027-04-22 (Estimated); Study Completion 2027-04-22 (Estimated)

PRIMARY OUTCOMES:
Time from study drug administration to complete cervical dilation | From study drug administration to complete cervical dilation, up to 24 hours.
  Time in hours from intravenous administration of papaverine or placebo after removal of the double-balloon catheter until complete cervical dilation (10 cm), as documented in the partogram/electronic medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Maor-Sagie, MD, Principal Investigator — Hillel Yaffe Medical Center; Rinat Gabbay-Benziv, Prof, Study Director — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: Undecided